CLINICAL TRIAL: NCT07108283
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Dose-Ranging Trial to Evaluate the Efficacy and Safety of Zasocitinib in Participants With Nonsegmental Vitiligo
Brief Title: A Study of Zasocitinib in Adults With Nonsegmental Vitiligo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-279-VT-2001; 2025-522309-40-00 (EU CTIS Number); jRCT2031250527 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-08-05; First posted 2025-08-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Nonsegmental Vitiligo
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Zasocitinib Low Dose (Experimental): Participants will receive Zasocitinib capsules, low dose, orally, up to Week 52.
  Interventions: Drug: Zasocitinib
- Zasocitinib Medium Dose (Experimental): Participants will receive Zasocitinib capsules, medium dose, orally, up to Week 52.
  Interventions: Drug: Zasocitinib
- Zasocitinib High Dose (Experimental): Participants will receive Zasocitinib capsules, high dose, orally, up to Week 52.
  Interventions: Drug: Zasocitinib
- Placebo Group 1/ Zasocitinib Medium Dose (Experimental): Participants will receive Placebo Group 1 orally, up to Week 24 followed by Zasocitinib capsules, medium dose, orally, up to Week 52.
  Interventions: Drug: Zasocitinib; Other: Placebo
- Placebo Group 2/ Zasocitinib High Dose (Experimental): Participants will receive Placebo Group 2, orally, up to Week 24 followed by Zasocitinib capsules, high dose, orally, up to Week 52.
  Interventions: Drug: Zasocitinib; Other: Placebo

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib capsules.
  Other Names: TAK-279
Other: Placebo — Zasocitinib matching placebo capsules.
  Arms: Placebo Group 1/ Zasocitinib Medium Dose; Placebo Group 2/ Zasocitinib High Dose

SUMMARY:
Vitiligo is a long-term autoimmune condition that causes the skin to lose its color. The body's germ-fighting system (immune system) mistakenly attacks the skin cells (melanocytes) which produce the pigment that gives the skin color (melanin). This leads to the formation of patches of skin with less or no pigment (depigmentation). These patches can occur anywhere on the body. In the nonsegmental form of vitiligo, similar patches occur on both sides of the body (symmetrical patches).

The main aim of this study is to learn how safe zasocitinib is, how well it works and how well it is tolerated by adults with nonsegmental vitiligo.

The participants will receive the study treatment (either zasocitinib or placebo) for up to 1 year (52 weeks). The placebo looks like the zasocitinib capsule but does not have any medicine in it. Participants who receive placebo at the beginning will change to zasocitinib after about 6 months.

During the study, participants will visit their study clinic 11 times.

ELIGIBILITY:
Inclusion criteria:

Participant willingness:

1. Participant is willing and able to understand and fully comply with trial procedures and requirements (including digital tools and applications), in the opinion of the investigator.
2. Participant has provided written informed consent and any required privacy authorization before the initiation of any trial procedures.

   Disease Characteristics:
3. Participants must have a clinical diagnosis of nonsegmental vitiligo: F-VASI greater than or equal to (>=) 0.5 and a T-VASI >= 5 and less than or equal to (<=) 50 at screening and Day 1.

   Age and Reproductive Status:
4. Participant is aged >=18 years to <=75 years old at the time of consent.
5. Participant meets the following birth control requirement:

   An individual with potential for pregnancy who is now of nonchildbearing potential with laboratory confirmation of postmenopausal status; or, if sexually active with a nonsterilized individual who produces sperm, an individual with potential for pregnancy who agrees to use a highly effective method of contraception from the signing of informed consent throughout the duration of the trial. The use of effective contraception will be required for assigned male sex at birth participants. In the European Union (EU) / European Economic Area (EEA) and the United Kingdom (UK), for participants who elect to use hormonal contraception as a form of highly effective contraception, the investigator must document a favorable benefit-risk assessment to justify the participant's inclusion in the trial at screening and every 3 months during the trial.
6. For participants in the EU/EEA or UK, the investigator must have no reason to believe that the participant would be placed at risk by participating in the trial with regard to the European Commission decision as of 10 March 2023 on measures to minimize risk of serious side effects with Janus Kinase inhibitor (JAKi) (EMA/142279/2023) and the UK MHRA guideline on JAKi: new measures to reduce risks of major cardiovascular events, malignancy, venous thromboembolism, serious infections and increased mortality as of 26 April 2023 (Drug Safety Update volume 16, issue 9).

Exclusion Criteria:

Target Disease-Related Exclusions:

1. Participant has segmental vitiligo.
2. Participant has >50 percent (%) leukotrichia on the face or >50% leukotrichia of the body (includes the face).
3. Participant requires immunomodulatory or immunosuppressive systemic treatment, other than nonsteroidal anti-inflammatory drugs, during the trial period for an immune-related disease (for example, inflammatory bowel disease).
4. Participant has a history of phototherapy (including, but not limited to, broadband Ultra-Violet [UV]-B, narrowband UV-B, psoralen and UV-A, excimer or other laser therapy, or tanning booth use) within 8 weeks before Day 1. Use of sunscreen products and protective apparel is recommended when sun exposure cannot be avoided.
5. Participant has concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the trial assessments.
6. History of any depigmenting or bleaching treatment for vitiligo or other skin disorder (for example, monobenzone or phenol).
7. History of any surgical treatments for vitiligo.
8. History of recent or progressive undiagnosed hearing loss.

   Recent/Concurrent Infectious Disease Exclusions:
9. Tuberculosis (TB):

   1. Participant has history of active TB infection, regardless of treatment status.
   2. Participant has signs or symptoms of active TB (including, but not limited to, chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator.
   3. Participant has evidence of Latent Tuberculosis Infection (LTBI) as evidenced by a positive QuantiFERON (QFT) result OR 2 indeterminate QFT results and participant does not have documentation of appropriate LTBI prophylaxis or is not able or not willing to initiate appropriate LTBI prophylaxis. Participant remains eligible if there are no signs/symptoms of active TB AND documentation of no history of active TB can be provided AND (1) participant can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines) or (2) participant has a positive QFT result or 2 indeterminate QFT results but has initiated prophylaxis (appropriate in duration and type per current local guidelines) a minimum of 2 weeks prior to Day 1. In the EU/ EEA and the UK, participants with evidence of LTBI, regardless of prophylaxis treatment status, must receive approval to participate in the trial from an infectious disease or other TB specialist (for example, pulmonologist).
   4. Participant has had any imaging trial during or 6 months prior to screening, including x-ray, chest Computed Tomography (CT), magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB. X-ray is required for all participants regardless of QuantiFERON-TB Gold results unless the participant has had normal chest imaging in the 6 months prior to screening. CT imaging is allowed per local sites requirements.
10. Herpes infections:

    1. Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1.
    2. Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
11. Non-herpetic viral diseases:

    1. Participant has presence of Hepatitis C Virus (HCV) antibody and a positive confirmatory test result for HCV Ribonucleic Acid (RNA) (nucleic acid test or polymerase chain reaction). In the EU/EEA and the UK, if the participant has total anti-HCV antibody positivity at screening but is confirmed to have no detectable HCV RNA by Polymerase Chain Reaction (PCR) testing, HCV RNA PCR testing will be assessed at additional visits per Schedule of Activities (SoA).
    2. Participant has presence of positive Hepatitis B surface antigen (HBsAg), or indeterminate HBsAg, presence of Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) (regardless of serology), or positive anti- Hepatitis B core antibody (HBcAb) without concurrent positive HBsAb. In the EU/EEA and the UK, if the participant has total anti-HBc antibody positivity at screening but is confirmed to have no detectable HBV DNA by PCR testing, the participant will repeat HBV DNA PCR testing at additional visits per SoA; if a participant has anti-HBsAb positivity at screening but is confirmed to have no detectable HBV DNA by PCR testing, unless the participant has documented completion of the HBV vaccination series by medical records, the participant will repeat HBV DNA PCR testing at additional visits per SoA. Note: For other countries in which there are hepatitis B screening guidelines, these can be done per local regulations or site's standard of care.
    3. Participant has positive results for Human Immunodeficiency Virus (HIV) by serology, regardless of viral load.
12. Other infectious diseases:

    1. Participant has a history of active infection or febrile illness within 7 days prior to Day 1, as assessed by the investigator.
    2. Participant has a history of symptoms suggestive of systemic or invasive infection within 30 days prior to Day 1.
    3. Participant has a history of bacterial, viral, or fungal infection that required hospitalization or treatment with intravenous antimicrobial therapy within 8 weeks prior to Day 1, or oral antimicrobial therapy within 30 days prior to Day 1.
    4. Participant has a history of chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial onychomycosis).
    5. Participant has a history of an infected joint prosthesis unless that prosthesis has been removed or replaced at least 60 days prior to Day 1.
    6. Participant has a history of opportunistic infections (for example, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
    7. Participant had a bacterial infection within 60 days prior to Day 1 for which he or she did not receive treatment.

    Noninfectious Disorders Exclusions:
13. Participant has any clinically significant medical condition, evidence of an unstable clinical condition (for example, cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, neurologic, nutritional, ophthalmologic or immunologic), or vital signs/physical/laboratory/Electrocardiogram (ECG) abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of trial results. These include but are not limited to:

    1. Participant has a history of known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
    2. Participant has a history of new or unstable autoimmune disease (including but not limited to thyroid disease, lupus, sjogrens, myasthenia gravis, or rheumatoid arthritis).
    3. Participant had a major surgery within 60 days prior to Day 1 or has a major surgery planned during the trial.
    4. Participant has unstable, poorly controlled, or severe hypertension at screening, confirmed by 2 repeat assessments.
    5. Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association criteria.
    6. Participant has a history of cancer or lymphoproliferative disease with the exception of successfully treated nonmetastatic cutaneous squamous cell carcinoma, basal cell carcinoma, or localized carcinoma in situ of the cervix. In the EU/EEA and the UK, for the participants with a history of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix, investigators must document a favorable benefit-risk assessment.
    7. For participants with asthma, chronic obstructive pulmonary disease, or other pulmonary illnesses has ever required intubation for treatment, currently requires oral corticosteroids, or has required more than 1 course of oral corticosteroids within 6 months prior to Day 1, or participant has been hospitalized within 3 months prior to Day 1.
    8. Participant has any of the following cardiovascular disease history:

       * A new diagnosis of atrial fibrillation or an episode of atrial fibrillation with rapid ventricular response or other dysrhythmia, non-acute cardiac hospitalization (for example, pacemaker implantation), pulmonary embolism, or deep venous thrombosis within the past 6 months prior to screening.
       * Any history of cerebrovascular event, myocardial infarction, coronary stenting, or aortocoronary bypass surgery. If, however, the investigator documents there are no suitable treatment alternatives available for the participant and it has been at least 6 months since the occurrence of any such event, the participant may enroll; in the EU/EEA and the UK, investigators must document a favorable benefit-risk assessment.
    9. Participant has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if they participated in the trial, in the opinion of the investigator.
    10. Participant has any lifetime history of suicide attempts, suicidal behavior, or active suicidal ideation with intent and plan based on medical history or a YES response to Columbia-Suicide Severity Rating Scale (C-SSRS) Questions 5; the participant has evidence of current active suicidal ideation based on YES response to questions 2, 3, 4, or 5 on C-SSRS Since Last Visit performed on Day1; or is clinically deemed to have a suicide risk by the investigator.
    11. Participant has a history of clinically significant drug or alcohol abuse within 12 months prior to Day 1.

    Laboratory/Physical Exclusions:
14. Participant has any of the following laboratory values at the screening visit:

    1. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) values >=3 times the Upper Limit of Normal (ULN).
    2. Total bilirubin (unconjugated and/or conjugated) ˃1.5 times the ULN.
    3. Hemoglobin (Hgb) <9.0 gram/deciliter (g/dL) (<90.0 gram/Liter [g/L]).
    4. Absolute white blood cell count less than (<) 3.0 * 10^9/Liter (L) (<3000/cubic millimeter [mm^3]).
    5. Absolute neutrophil count of <1.0 * 10^9/L (<1000/mm^3).
    6. Absolute lymphocyte count of <0.5 * 10^9/L (<500/mm^3).
    7. Platelet count <100 * 10^9/L (<100,000/mm^3).
    8. Thyroid Stimulating Hormone (TSH) outside the normal reference range AND free T4 or T3 outside the normal reference range.
    9. Estimated creatinine clearance <30 milliliter/minute (mL/min) based on the Cockcroft-Gault calculation.
    10. Creatine Phosphokinase (CPK) > ULN. CPK may be repeated once; if repeat value is Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or lower (or <=2.5 × ULN) and no higher than the initial value, participant remains eligible. Investigators should assess the participant for modulating factors including concomitant medications or vigorous exercise that may affect CPK levels.
15. Participant has any other significant laboratory abnormalities that, in the opinion of the investigator, might place the participant at unacceptable risk for participation in this trial.
16. Participant does not tolerate venipuncture or inability to be venipunctured.

    Allergies and Adverse Drug Reactions Exclusions:
17. Participant has a history of significant drug allergy (such as anaphylaxis).
18. Participant has a known or suspected allergy to zasocitinib or any of its components.

    Other Exclusions:
19. Participant has a positive pregnancy test result or plans to become pregnant during the trial period, including plans to undergo in vitro fertilization, donate ova (eggs), or sperm, or participant is lactating/nursing.
20. Participant has given greater than 500 mL of blood or plasma within 30 days of screening (during a clinical trial or at a blood bank donation) or plans to donate blood during the course of the trial.
21. Participant is compulsorily detained for treatment of either a psychiatric or physical (for example, infectious disease) illness, or is committed to an institution (for example, prison) by virtue of an order issued either by judicial or administrative authorities.
22. Participant is a trial site employee, an immediate family member (for example, spouse, parent, child, sibling), or is in a dependent relationship with trial site employee who is involved in the conduct of this trial or may consent under duress.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-10-12 (Estimated); Study Completion 2027-11-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving >= 75% Improvement From Baseline in Facial Vitiligo Area Scoring Index (F-VASI) at Week 24 | Baseline, Week 24
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.5, with higher scores indicating more severe disease. Negative changes from baseline indicate improvement. This is recorded as either Yes (achieved >= 75% improvement) or No (did not achieve).

SECONDARY OUTCOMES:
Percent Change From Baseline in the F-VASI at Week 24 | Baseline, Week 24
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.5, with higher scores indicating more severe disease. Negative changes from baseline indicate improvement.
Percent Change From Baseline in the Total- Vitiligo Area Scoring Index (T-VASI) at Week 24 | Baseline, Week 24
  The VASI is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100, with higher scores indicating more severe disease.
Percentage of Participants Achieving F-VASI 50 at Week 24 | At Week 24
  F-VASI 50 is defined as >=50% improvement from baseline.
Percentage of Participants Achieving T-VASI 50 at Week 24 | At Week 24
  T-VASI 50 is defined as >=50% improvement from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (70):
- United States (23):
  - Dermatology Trial Associates, Bryant, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - The Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - UC Davis Department of Dermatology, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - Encore Medical Research of Boynton Beach LLC., Boynton Beach, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Advanced Clinical Research Institute (ACRI), Tampa, Florida
  - Encore Medical Research of Weston LLC, Weston, Florida
  - DelRicht Research - Dermatology, Baton Rouge, Louisiana
  - DelRicht Research (Audubon Dermatology), New Orleans, Louisiana
  - Lawrence J Green LLC, Rockville, Maryland
  - Hamzavi Dermatology - Canton, Canton, Michigan
  - Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Markowitz Medical dba Optiskin, New York, New York
  - Bexley Dermatology (legal entity - Dermatologists of Southwestern Ohio, LLC), Bexley, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Health Science Center Houston, Bellaire, Texas
  - ACRC Trials, Plano, Texas
  - Progressive Clinical Research-San Antonio, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Canada (8):
  - Brunswick Dermatology Center (BDC), Fredericton, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - LEADER research, Hamilton, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - North York Research Inc, Toronto, Ontario
  - Centre de Recherche Dermatologique de Quebec, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- China (5):
  - The First Hospital of Wuhan, Wuhan, Hubei
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
- France (6):
  - Bordeaux University Hospital, Bordeaux
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopitaux Universitaires Henri Mondor (Hopital Henri-Mondor), Créteil
  - Centre Hospitalier Le Mans (CHM), Le Mans
  - Cabinet Médical du Dr Ruer, Martigues
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital Larrey, Toulouse
- Italy (5):
  - Humanitas Research Hospital, Rozzano, Milan
  - Istituto Dermopatico Immacolata IDI, IRCCS, Rome, Roma
  - Spedali Civili Hospital, Brescia
  - Azienda Usl Toscana Centro, Florence
  - Fondazione Policlinico A. Gemelli, Rome
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toho University-Sakura Hospital Medical Center, Sakura-shi, Chiba
  - Kume Clinic - Sakai, Nishi-ku, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Mexico (4):
  - CRI Centro Regiomontano de Investigation SC, Monterrey, New Leon
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Clinica de Enfermedades Cronicas y de Procedimientos Especiales, Morelia, Predeterminado
  - Arke SMO SA de CV, Veracruz
- Poland (8):
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski, Osielsko, Kuyavian-Pomeranian Voivodeship
  - dermMedica Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Szczecińskie Centrum Medyczne Sp. z o.o., Szczecin, West Pomeranian Voivodeship
  - Gyncentrum Sp. z o.o., Katowice
  - Klinika Dermatologii i Dermatologii Onkologicznej Uniw. Szp. Klin. in Rzeszów, Rzeszów
  - ETG Warszawa, Warsaw
  - Dermoklinika Centrum Medyczne, Lodz, Łódź Voivodeship
  - Dermedic Jacek Zdybski, Kielce, Świętokrzyskie Voivodeship
- Spain (6):
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario La Paz (HULP), Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital de Manises, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/9d9c2ce1337c4adc??page=1&idFilter=TAK-279-VT-2001